CLINICAL TRIAL: NCT03218215
Title: Physiological Study About Advantages of Monitoring Mechanical Assisted Cough
Brief Title: Monitoring Mechanical Assisted Cough
Acronym: MONICA
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Fundacio Catalana de Pneumologia (Other)
Responsible Party: Principal Investigator, Cristina Lalmolda-Puyol, Physiotherapist, Corporacion Parc Tauli
Other Study IDs: SOCAP-2015
Record Dates: First submitted 2017-07-07; First posted 2017-07-14 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Neuromuscular Diseases; Respiratory Complication
Keywords: cough assits
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Mechanical assistance cough for patients with neuromuscular disorders (NMD) are known, but there is no adaptation model established. Currently is performed subjectively by the physiotherapist following the pressures recommended in the current literature as optimal (±40CmH2O). To check is these pressures are the most optimal pressures to achieve the better peak cough flow (PCF) monitoring cough assist (Mechanical insuffllation-exsuflattion MI-E) maneuvers and analyzing pressure- flow / time curves

Adults with MI-E criteria (PCFbaseline <160 l /min). A pneumotachograph, PeakAnalysis software and nasobucal mask were used to monitor and analyze flow/time curves. Protocol included 9 PCF values in each patient: 1 baseline, 4 related with inspiratory pressure in sequential increase of 10 cmH2O (10 to 40 cmH2O) and 4 adding expiratory pressures (±10 to ±40cmH2O)

DETAILED DESCRIPTION:
A cross-sectional observational study was performed with patients with NMD who had PFC below 160l/min according to Mechanical insufflation- exsufflation (MI-E ) criteria to assit the cough.

Exclusion criteria were age <18 years, patients who had undergone tracheostomy, exacerbated or with psychiatric problems and patients with relative contraindications (bullous emphysema background, risk of pneumothorax or recent barotrauma).

MI- E study protocol An original protocol was established to perform treatment assessment with Cough Assitst T70 MI-E device® Phillips Respironics. Protocol based on 9 phases of monitoring cough. First was baseline performed for the patient without mechanical assistance and the others were performed by incremental inspiratory and expiratory pressures (cm H2O). Considering ±40 cmH2O as optimal, it was the maximum at the study. An increase of 10 cm H2O in each phase was made starting with the inspiratory pressure (10 to 40 cm H2O or maximum tolerated). Once the maximum pressure tolerated by the patient was reached, the expiratory pressure was introduced following the same sequence. (-10 to -40 cm H2O or maximum tolerated).

Monitoring MI- E protocol: signals and instrumentation As a signal acquisition system, an external polygraph (16Sp Powerlab, ADInstruments, Sydney, Australia), equipped with a pressure transducer (1050 model) and a pneumotachograph (S300, instrumental dead space _ 70 mL, resistance _ 0.0018 cm H2O/L/s) was connected to MI-E device. Sampling frequency was set to 200 Hz, and the polygraph was connected to a personal computer equipped with Chart 7.0 software for Windows.

Signal processing and analysis of waveforms, pressure-time and flow-time, were performed by this software that allowed calculate Peak cough flow maximum in each phase and checking possible respiratory events what could happen during the therapy.

Parameters measured and Other assessments PCFMaximal (max) (l /min) achieved by the patient measured thorough Peak Analysis software, related to Maximal Inspiratory pressure (MIP) and Maximal Expiratory pressure (MEP) measured by cmH2O, and Phase Number like a combination of both outcomes. All phases recorded 3 respiratory cycles with cough and the best was used for the analysis.

Oxygen saturation (SpO2%)and heart rate (bpm), before and after of each phase to control patient status. Patients with Amyotrophic Lateral Sclerosis (ALS) were assessed using th ALS Functional Rating Scale revised (ALSFRS-r) (cita). Bulbar impairment score was evaluated from the ALSFRS-r, from where the items of speech and swallowing were calculated.

ELIGIBILITY:
Inclusion Criteria:

* patients with NMD who had PFC below 160l/min according to Mechanical insufflation- exsufflation (MI-E ) criteria to assit the cough.

Exclusion Criteria:

* age <18 years,
* patients who had undergone tracheostomy, exacerbated or with psychiatric problems
* patients with relative contraindications (bullous emphysema background, risk of pneumothorax or recent barotrauma).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with NMD who had PFC below 160l/min according to Mechanical insufflation- exsufflation (MI-E ) criteria to assit the cough.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-05-26 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Peak cough flow (max): PCFmax (l/min) | Day 1
  Peak cough flow maximum achieve by the patient. This outcome will be related with outcomes pressures.
Max Inspiratory Pressure: MIP (cmH2O) | Day 1
  Inspiratory pressure in phase of protocol with the best peak cough flow achieve
Max Expiratory Pressure:MEP (cmH2O) | Day 1
  Expiratory pressure in phase of protocol with the best peak cough flow achieve

SECONDARY OUTCOMES:
Oxygen Saturation pre protocol | Day 1
  Oxygen saturation pre protocol measured by %
Oxygen Saturation post protocol | Day 1
  Oxygen saturation post protocol measured by %
ALSFR scale | Day 1
  scale that measure level of disease progression in ALS ( amiotrophic Lateral Sclerosis) main pathology of study
Pathology | Day 1
  ALS, other neumuscular disorders
PCF at baseline (l/min) | Day 1
  PCF achieve before the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Manel Lujan, MD, Study Director — Corporacion Parc Tauli